CLINICAL TRIAL: NCT06364670
Title: Application of Machine Learning Based on fNIRS in Predicting Acupuncture's Efficacy in Treating Tinnitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Hantong Hu, M.D., The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSLL-KY-2023-011-01
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Tinnitus
Keywords: acupuncture; moxibustion; tinnitus; fNIRS; machine learning
MeSH Terms: conditions — Tinnitus | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The acupuncture group (Experimental): Subjects in the acupuncture group will undergo acupuncture treatment, which is administered 3 times a week for 4 weeks.
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture — Acupuncture will be performed at acupoints including TE17 (Yifeng), SI19 (Tinggong), GB2 (Tinghui), TE5 (Waiguan), TE3 (Zhongzhu), ST36 (Zusanli ), KI3 (Taixi), and etc.

SUMMARY:
This trial aims to use machine learning to analyze fNIRS imaging data of specific brain regions of tinnitus patients, thereby constructing a predictive model of the clinical efficacy of acupuncture for SNT.

DETAILED DESCRIPTION:
This study will recruit 500 subjects with tinnitus. Functional near-infrared spectroscopy (fNIRS) will be employed to examine specific brain regions, and the corresponding fNIRS imaging data from all detection channels will be extracted. Subsequently, the subjects will undergo a course of acupuncture treatment. Based on the recovery status of tinnitus at the conclusion of the acupuncture course, all subjects will be categorized into a "good prognosis group" and a "poor prognosis group" according to relevant efficacy criteria. The entire dataset will then be randomly divided into a training set (70%) and a test set (30%) following a 7:3 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral tinnitus that meets the diagnostic criteria for chronic subjective tinnitus.
* Male and female, aged between 18 and 60 years.
* Right-handed subjects who are able to comply with the study protocol and sign written informed consent.
* Not participating in other clinical trials concurrently.

Exclusion Criteria:

* Participants with objective tinnitus.
* Participants have nervous system diseases or neuropsychiatric diseases that can significantly affect brain blood oxygen metabolism assessed by fNIRS.
* Participants with severe cardiovascular and cerebrovascular diseases, malignant liver and kidney diseases, and other serious diseases.
* Participants have any contraindications for acupuncture (such as a bleeding tendency).
* Pregnant or lactating women.
* Participants have received tinnitus treatment with drugs or other therapies in the last four weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in resting-state functional connectivity (RSFC) | at baseline (pre-treatment), after 4-week treatment
  RSFC will be measured by functional near-infrared spectroscopy (fNIRS).
Change in hemoglobin signals | at baseline (pre-treatment), after 4-week treatment
  Hemoglobin signals will be measured by functional near-infrared spectroscopy (fNIRS).
Change in Tinnitus Severity Grading | at baseline (pre-treatment), after 4-week treatment
  Tinnitus Severity Grading is based on relevant expert consensus.

SECONDARY OUTCOMES:
Change in Tinnitus Handicap Inventory score | at baseline (pre-treatment), after 4-week treatment
  Tinnitus Handicap Inventory contains 25 items, each valued at 0-4 points. A larger score indicates a more severe degree of tinnitus.
Change in average pure-tone threshold | at baseline (pre-treatment), after 4-week treatment
  The average pure-tone threshold will be assessed by pure-tone audiometry.

CONTACTS AND LOCATIONS:
Overall Officials: Hantong Hu, M.D, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- the Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang X, Jiang D, Kong D, Liu H, Chen L, Li Y, Zhou J, Gao H, Hu H. Predicting Individual Response to Acupuncture in Sensorineural Tinnitus Using Integrated Functional Near-Infrared Spectroscopy and Machine Learning: Protocol for a Model Development and Validation Study. J Multidiscip Healthc. 2025 Oct 9;18:6579-6593. doi: 10.2147/JMDH.S550296. eCollection 2025. PMID 41089742